CLINICAL TRIAL: NCT03671759
Title: Coffee and Real-time Atrial and Ventricular Ectopy
Acronym: CRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-25195
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Premature Atrial Contractions; Premature Ventricular Contractions
Keywords: Caffeine; Coffee; Arrhythmias; Palpitations; Cardiac ectopy; PACs; PVCs
MeSH Terms: conditions — Atrial Premature Complexes; Ventricular Premature Complexes; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: N-of-1 (Experimental): Participants will be randomized in two-day blocks to consume then avoid caffeine ("Start: On Caffeine") or avoid then consume caffeine ("Start: Off Caffeine"). Using an N-of-1 strategy delivered by the NIH-funded, UCSF-run Eureka platform utilizing a mobile smartphone-based application, participants will receive instructions and answer questions to help us understand the relationship between caffeine and heart rhythm.
  Interventions: Behavioral: Start: On Caffeine; Behavioral: Start: Off Caffeine

INTERVENTIONS:
Behavioral: Start: On Caffeine — In this two-day block, participants will be instructed to consume caffeine for one day and avoid caffeine the next day.
Behavioral: Start: Off Caffeine — In this two-day block, participants will be instructed to avoid caffeine for one day and consume caffeine the next day.

SUMMARY:
Atrial fibrillation (AF) and heart failure (HF) are morbid, costly, and incompletely understood diseases that have reached epidemic proportions worldwide. A dose-dependent relationship exists between premature atrial and ventricular contractions (PACs and PVCs) and development of AF and HF, respectively. Identifying and understanding the mechanisms of additional modifiable risk factors for ectopy has the potential to markedly reduce the healthcare burden of these diseases. In considering how to modify the prevalence of these ectopic beats, the investigators believe common exposures in daily life are prime candidates. Current guidelines suggest that caffeine may be an important trigger for frequent ectopy, although large population-based studies have not demonstrated an association between caffeine consumption and development of clinically significant arrhythmias. No study has employed an actual randomization intervention to assess the effects of caffeine on cardiac ectopy. Utilizing the Eureka platform, the investigators plan to utilize the N-of-1 strategy to rigorously investigate the real-time effect of caffeine intake on ectopy.

DETAILED DESCRIPTION:
This study is designed as a N to 1 randomized trial, where each participant will be randomized to consume or abstain from coffee each day of a 14 day monitoring period. Participants will wear an automatically recording electrocardiographic monitor (ZIO® XT Patch), continuous glucose monitor (Dexcom G6), and a fitness tracker (Fitbit INSPIRE) while utilizing Eureka-a mobile application. We will compare participant self-report of caffeine consumption, glucose monitoring, fitness levels, sleep health, and heart rhythm data in order to better understand the relationship between acute caffeine consumption and heart rhythm changes. Participants will also be genotyped for caffeine metabolism-related SNPs. A total of 100 participants will be enrolled at the UCSF study site.

ELIGIBILITY:
Inclusion Criteria:

1. Are age 18 or older
2. Have a smartphone
3. Are able to use the Eureka mobile application
4. Are willing to provide a saliva sample for genetic processing
5. Drink coffee or coffee-based products at least once a year
6. Are willing to abstain from coffee, caffeinated products, or minimally caffeinated products (decaffeinated coffee) for at least 2 days when instructed

Exclusion Criteria:

1. Have a history of atrial fibrillation, heart failure
2. Have an ICD or pacemaker
3. Have treatment with beta blockers, non-dihydropyridine calcium channel blockers, or Vaughn-Williams class 1 or 3 antiarrhythmic medications
4. Have a medical reason to avoid coffee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Change in PAC frequency | Baseline and after completion of coffee consumption, up to 2 weeks
  Participants will be wearing a continuously recording ECG monitor for two weeks. The primary outcome will be change in premature atrial contraction (PAC) frequency due to caffeine consumption or avoidance during the enrollment period.

SECONDARY OUTCOMES:
Change in SVT episodes | Baseline and after completion of coffee consumption, up to 2 weeks
  Participants will be wearing a continuously recording ECG monitor for two weeks. A secondary outcome will be change in supraventricular tachycardia (SVT) episodes due to caffeine consumption or avoidance during the enrollment period.
Change in VT episodes | Baseline and after completion of coffee consumption, up to 2 weeks
  Participants will be wearing a continuously recording ECG monitor for two weeks. A secondary outcome will be change in ventricular tachycardia (VT) episodes episodes due to caffeine consumption or avoidance during the enrollment period.
Mean daily glucose levels | 2 weeks
  Participants will be wearing a continuous glucose monitor (Dexcom G6) that will record serum glucose levels. A secondary outcome will be difference in mean daily glucose levels due to caffeine consumption or avoidance during the enrollment period.
Mean step count | 2 weeks
  Participants will be wearing a fitness tracker (Fitbit INSPIRE) that will record step counts. A secondary outcome will be difference in mean step counts due to caffeine consumption or avoidance during the enrollment period.
Mean sleep duration | 2 weeks
  Participants will be wearing a fitness tracker (Fitbit INSPIRE) that will record sleep duration. A secondary outcome will be difference in mean sleep duration due to caffeine consumption or avoidance during the enrollment period.
Change in PVC frequency | Baseline and after completion of coffee consumption, up to 2 weeks
  Participants will be wearing a continuously recording ECG monitor for two weeks. The primary outcome will be change in ventricular contraction (PVC) frequency due to caffeine consumption or avoidance during the enrollment period.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Marcus, MD, MAS, Principal Investigator — University of California, San Francisco; David Rosenthal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chugh SS, Blackshear JL, Shen WK, Hammill SC, Gersh BJ. Epidemiology and natural history of atrial fibrillation: clinical implications. J Am Coll Cardiol. 2001 Feb;37(2):371-8. doi: 10.1016/s0735-1097(00)01107-4. PMID 11216949
- [Background] Coyne KS, Paramore C, Grandy S, Mercader M, Reynolds M, Zimetbaum P. Assessing the direct costs of treating nonvalvular atrial fibrillation in the United States. Value Health. 2006 Sep-Oct;9(5):348-56. doi: 10.1111/j.1524-4733.2006.00124.x. PMID 16961553
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Dewland TA, Vittinghoff E, Mandyam MC, Heckbert SR, Siscovick DS, Stein PK, Psaty BM, Sotoodehnia N, Gottdiener JS, Marcus GM. Atrial ectopy as a predictor of incident atrial fibrillation: a cohort study. Ann Intern Med. 2013 Dec 3;159(11):721-8. doi: 10.7326/0003-4819-159-11-201312030-00004. PMID 24297188
- [Background] Dukes JW, Dewland TA, Vittinghoff E, Mandyam MC, Heckbert SR, Siscovick DS, Stein PK, Psaty BM, Sotoodehnia N, Gottdiener JS, Marcus GM. Ventricular Ectopy as a Predictor of Heart Failure and Death. J Am Coll Cardiol. 2015 Jul 14;66(2):101-9. doi: 10.1016/j.jacc.2015.04.062. PMID 26160626
- [Background] Blomstrom-Lundqvist C, Scheinman MM, Aliot EM, Alpert JS, Calkins H, Camm AJ, Campbell WB, Haines DE, Kuck KH, Lerman BB, Miller DD, Shaeffer CW, Stevenson WG, Tomaselli GF, Antman EM, Smith SC Jr, Alpert JS, Faxon DP, Fuster V, Gibbons RJ, Gregoratos G, Hiratzka LF, Hunt SA, Jacobs AK, Russell RO Jr, Priori SG, Blanc JJ, Budaj A, Burgos EF, Cowie M, Deckers JW, Garcia MA, Klein WW, Lekakis J, Lindahl B, Mazzotta G, Morais JC, Oto A, Smiseth O, Trappe HJ; European Society of Cardiology Committee, NASPE-Heart Rhythm Society. ACC/AHA/ESC guidelines for the management of patients with supraventricular arrhythmias--executive summary. a report of the American college of cardiology/American heart association task force on practice guidelines and the European society of cardiology committee for practice guidelines (writing committee to develop guidelines for the management of patients with supraventricular arrhythmias) developed in collaboration with NASPE-Heart Rhythm Society. J Am Coll Cardiol. 2003 Oct 15;42(8):1493-531. doi: 10.1016/j.jacc.2003.08.013. No abstract available. PMID 14563598
- [Background] Dixit S, Stein PK, Dewland TA, Dukes JW, Vittinghoff E, Heckbert SR, Marcus GM. Consumption of Caffeinated Products and Cardiac Ectopy. J Am Heart Assoc. 2016 Jan 26;5(1):e002503. doi: 10.1161/JAHA.115.002503. PMID 26813889
- [Derived] Marcus GM, Rosenthal DG, Nah G, Vittinghoff E, Fang C, Ogomori K, Joyce S, Yilmaz D, Yang V, Kessedjian T, Wilson E, Yang M, Chang K, Wall G, Olgin JE. Acute Effects of Coffee Consumption on Health among Ambulatory Adults. N Engl J Med. 2023 Mar 23;388(12):1092-1100. doi: 10.1056/NEJMoa2204737. PMID 36947466
- See also: Ventricular Premature Complexes Treatment & Management — http://emedicine.medscape.com/article/158939-treatment-a1130